CLINICAL TRIAL: NCT04023812
Title: Real-World Molecular Testing, Treatment Patterns and Clinical Outcomes in Chinese Patients With Stage III NSCLC- A Prospective, Non-Interventional Study(MOOREA)
Brief Title: Stage III NSCLC RWE in Chinese Patients
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D4194R00009
Record Dates: First submitted 2019-05-30; First posted 2019-07-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: prospective; observational; stage III NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Cohort 1, including patients without surgical resection, will be defined as unresectable stage III NSCLC
- Cohort 2: Cohort 2,including patients with surgical resection, will be defined as resectable stage III NSCLC

SUMMARY:
The objectives of this study are to assess molecular testing, treatment patterns and associated clinical outcomes in Chinese patients with treatment-naïve stage III non-small cell lung cancer (NSCLC) in real world setting. This study is a prospective, non-interventional study. It is descriptive in nature and does not attempt to test any specific a priori hypotheses.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 years or older.
* Provision of informed consent prior to any study specific procedures.
* Histologically or cytologically confirmed locally advanced, stage III NSCLC (according to version 8 of the International Association for the Study of Lung Cancer Staging Manual in Thoracic Oncology; IASLC Staging Manual in Thoracic Oncology).

Exclusion Criteria:

* Enrolment in studies that prohibit any participation in this observational study.

  * Patients may be concurrently enrolled in unblinded clinical trials, but not blinded clinical trials in which the treatment being administered is unknown.
* Prior surgery, radiotherapy or systemic therapy for NSCLC, including chemotherapy, targeted therapy, anti-angiogenesis, etc.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stage III NSCLC patients who received no prior systemic therapy for NSCLC before study enrolment
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2019-07-16 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
To observe treatment patterns of unresectable, stage III NSCLC | Date of enrollment in the study until end of follow-up or death if this occurs before, assessed approximately up to 36 months
  Treatment received before disease progress including chemotherapy, targeted therapy, immunotherapy, anti-angiogenesis therapy and radiotherapy

SECONDARY OUTCOMES:
To observe the clinical outcome of unresectable, stage III NSCLC | Date of enrollment in the study until end of follow-up or death if this occurs before, assessed approximately up to 36 months
  Overall survival measured from the date of treatment initiation in the study to the date of death due to any cause; Progression-free Survival (PFS) measured from the date of treatment initiation in the study, until physician-reported progression or death due to any cause, whichever occurs first.
To observe molecular testing patterns of stage III NSCLC | Date of enrollment in the study until end of follow-up or death if this occurs before, assessed approximately up to 36 months
  Molecular testing patterns including:
  Molecular testing rate defined as the number of patients who received molecular testing divided by total patient's number; Molecular testing details including sample type, test type; Molecular testing results.
To estimate parameters associated with radiation pneumonitis | Date of enrollment in the study until end of follow-up or death if this occurs before, assessed approximately up to 36 months
  Assessment of radiation pneumonitis observed with radiotherapy among patients with unresectable, stage III NSCLC
To observe adjuvant treatment patterns of resectable, stage III NSCLC | Date of enrollment in the study until end of follow-up or death if this occurs before, assessed approximately up to 36 months
  Adjuvant treatment received post surgery including chemotherapy, targeted therapy and radiotherapy.

CONTACTS AND LOCATIONS:
Locations (17):
- China (17):
  - Research Site, Beijing, China
  - Research Site, Datong, China
  - Research Site, Fenyang, China
  - Research Site, Guangzhou, China
  - Research Site, Hefei, China
  - Research Site, Jinan, China
  - Research Site, Nanning, China
  - Research Site, Qingdao, China
  - Research Site, Shantou, China
  - Research Site, Taizhou, China
  - Research Site, Tianjin, China
  - Research Site, Yinchuan, China
  - Research Site, Changchun
  - Research Site, Chengdu
  - Research Site, Hong Kong
  - Research Site, Shanghai
  - Research Site, Shijiazhuang

REFERENCES:
- See also: CSR Synopsis_redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D4194R00009&attachmentIdentifier=c7e1a4f3-4549-4081-9e14-53866eee2062&fileName=Moorea-Clinical_Study_Report_Synopsis.pdf&versionIdentifier=